CLINICAL TRIAL: NCT01769586
Title: Randomized Trial of Diphenhydramine Versus Continued Midazolam in "Difficult-to-sedate" Patients Undergoing Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0003
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Sedation; Endoscopy
Keywords: Sedation; Endoscopy; Diphenhydramine; Midazolam
MeSH Terms: interventions — Diphenhydramine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diphenhydramine (Active Comparator): Increments of 25 mcg to maximum of 3 times (total 75 mcg)
  Interventions: Drug: Diphenhydramine
- Midazolam (Active Comparator): 1.5 mg increments up to 3 times (maximum 4.5 mg)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Diphenhydramine
  Arms: Diphenhydramine
Drug: Midazolam
  Arms: Midazolam

SUMMARY:
Patients who are undergoing colonoscopy and are not adequately sedated after initial standard sedation with midazolam 5 mg and fentanyl 100 mcg will be randomly assigned to receive diphenhydramine vs. continued midazolam, and their level of sedation will be assessed. Our hypothesis is that diphenhydramine will provide better sedation than continued administration of midazolam during colonoscopy in patients not achieving adequate sedation with standard doses of midazolam plus fentanyl.

DETAILED DESCRIPTION:
Patients who are undergoing colonoscopy and are not adequately sedated after initial standard sedation with midazolam 5 mg and fentanyl 100 mcg will be randomly assigned to receive diphenhydramine (up to 3 incremental doses of 25 mcg each) vs. continued midazolam (up to 3 incremental doses of 1.5 mg each). the level of sedation will be assessed using the MOAA/S scale 2-3 minutes after each administration to determine if they are sufficiently sedated to begin colonoscopy. The patient, the healthcare team involved in performing the endoscopy, and the investigator assessing sedation will be blinded to the therapy. Our hypothesis is that diphenhydramine will provide better sedation than continued administration of midazolam during colonoscopy in patients not achieving adequate sedation with standard doses of midazolam plus fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years-old who are undergoing elective colonoscopy with conscious sedation

Exclusion Criteria:

* allergy or prior adverse reactions to diphenhydramine
* medical contraindications to use of diphenhydramine (e.g. closed angle glaucoma)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loren Laine, MD, Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Sachar H, Pichetshote N, Nandigam K, Vaidya K, Laine L. Continued midazolam versus diphenhydramine in difficult-to-sedate patients: a randomized double-blind trial. Gastrointest Endosc. 2018 May;87(5):1297-1303. doi: 10.1016/j.gie.2017.01.028. Epub 2017 Jan 31. PMID 28159539

RESULTS

PARTICIPANT FLOW:
Groups:
- Diphenhydramine: Increments of 25 mcg to maximum of 3 times (total 75 mcg)
  Diphenhydramine
- Midazolam: 1.5 mg increments up to 3 times (maximum 4.5 mg)
  Midazolam
Period: Overall Study
Arm/Group | Diphenhydramine | Midazolam
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diphenhydramine | Midazolam | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Full Range); unit: years] | 60 [28 to 76] | 61 [27 to 76] | 60 [27 to 76]
Gender [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 94 | 93 | 187

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieve Adequate Sedation to Allow Colonoscopy (Defined as MOAA/S ≤3)
Description: Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scale. This scale ranges from 0 to 5, where 0 denotes general anesthesia, in which the patient has no response to painful stimuli, and 5 denotes a level of minimal sedation in which the patient is fully awake.
Time Frame: Approximately 10 minutes or less
Measure: Number; unit: participants
Arm/Group | Diphenhydramine | Midazolam
Number analyzed (Participants) | 100 | 100
participants | 27 | 65
Statistical Analysis 1: Comparison: Diphenhydramine vs Midazolam; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Difference (RD) = .38, 95% CI 2-sided [.24 to .50]

ADVERSE EVENTS:
Arm/Group | Diphenhydramine | Midazolam
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 2/100 | 8/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diphenhydramine (N=100) | Midazolam (N=100)
Desaturation (General disorders) | 1 | 2
Hypotension (General disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes